CLINICAL TRIAL: NCT00774332
Title: A Phase II Study of CODOX-M/ IVAC in Relapsed/Refractory ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: Yeungnam University College of Medicine, Yeungnam University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-011
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ANAVACYM protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CODOX-M — Cytoxan,Mesna,Adriamycin,Vincristine,Methotrexate,Leucovorin,Cytarabine

SUMMARY:
A Phase II Study of CODOX-M/ IVAC in Relapsed/Refractory ALL

DETAILED DESCRIPTION:
The feasibility will be evaluated in terms of complete remission rate, duration of complete remission, disease-free survival, overall survival, and toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/resistant acute lymphoblastic leukemia
* Patients must be between 15 and 65 years of age.
* Estimated life expectancy of more than 3 months
* ECOG performance status of 2 or lower, Karnofsky scale > 60 (see appendix I)
* Adequate cardiac function (EF>45%) on echocardiogram or MUGA scan
* Adequate kidney function (estimated Ccr >50 ml/min)

Exclusion Criteria:

* Patients with CNS involvement of leukemic blasts will not be excluded.
* Patients with extramedullary relapse(s) only will be excluded.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2006-06; Primary Completion 2006-06 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Duration of complete remission, disease-free survival, overall survival, toxicities | 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Hee Lee, Doctor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea